CLINICAL TRIAL: NCT07129993
Title: A Randomized, Open-Label, Phase 2/3 Study of Datopotamab Deruxtecan (Dato-DXd) Plus Carboplatin or Cisplatin Versus Gemcitabine Plus Carboplatin or Cisplatin in Participants With Locally Advanced or Metastatic Urothelial Carcinoma (la/mUC) Who Progressed During or After Enfortumab Vedotin (EV) Plus Pembrolizumab Combination Treatment TROPION-Urothelial03 (TU03)
Brief Title: Study of Datopotamab Deruxtecan Plus Carboplatin or Cisplatin Versus Gemcitabine Plus Carboplatin or Cisplatin in Participants With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-328
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Urothelial Cancer; Bladder Cancer
Keywords: Urothelial Carcinoma; Dato-DXd; TROPION; DS-1062a; Datopotamab Deruxtecan
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Carboplatin; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Phase 2): Dato-DXd, 4 mg/kg with Platinum (Experimental): Participants will receive Dato-DXd in combination with platinum (carboplatin or cisplatin). The RP3D will be determined using data collected from Part A.
  Interventions: Drug: Dato-DXd; Drug: Carboplatin; Drug: Cisplatin
- Part A (Phase 2): Dato-DXd, 6 mg/kg with Platinum (Experimental): Participants will receive Dato-DXd in combination with platinum (carboplatin or cisplatin). The RP3D will be determined using data collected from Part A.
  Interventions: Drug: Dato-DXd; Drug: Carboplatin; Drug: Cisplatin
- Part B (Phase 3): Dato-DXd, RP3D with Platinum (Experimental): Participants will receive Dato-DXd at the RP3D in combination with platinum (carboplatin or cisplatin).
  Interventions: Drug: Dato-DXd; Drug: Carboplatin; Drug: Cisplatin
- Part B (Phase 3): Gemcitabine with Platinum (Active Comparator): Participants will receive Gemcitabine in combination with platinum (carboplatin or cisplatin).
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Dato-DXd — Dato-DXd will be administered as an intravenous (IV) infusion every three weeks (Q3W) at a dose of 4 mg/kg or 6 mg/kg in Part A or RP3D in Part B
  Other Names: Datopotamab Deruxtecan
  Arms: Part A (Phase 2): Dato-DXd, 4 mg/kg with Platinum; Part A (Phase 2): Dato-DXd, 6 mg/kg with Platinum; Part B (Phase 3): Dato-DXd, RP3D with Platinum
Drug: Carboplatin — Carboplatin will be administered as an intravenous (IV) infusion every three weeks (Q3W) at a dose of AUC 4.5 or 5.0 mg•min/mL
Drug: Cisplatin — Cisplatin will be administered as an intravenous (IV) infusion every three weeks (Q3W) at a dose of 70 mg/m2
Drug: Gemcitabine — Gemcitabine will be administered as an IV infusion at a dose of 1000 mg/m2 on Day 1 and 8 of every 3 week cycle.
  Arms: Part B (Phase 3): Gemcitabine with Platinum

SUMMARY:
This is a global, multicenter, randomized, open-label, Phase 2/3 study of Dato-DXd plus carboplatin or cisplatin versus gemcitabine plus carboplatin or cisplatin in participants with la/mUC who progressed during or after EV plus pembrolizumab combination treatment.

This trial will start with part A, Phase 2. During part A, Phase 2, preliminary efficacy and safety will be assessed, and the recommended Phase 3 dose (RP3D) will be identified when the data allow sufficient assessment of activity, safety, and tolerability. The Phase 3 part will start contingent upon the assessment in the Phase 2 part, taking into consideration the totality of information.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult ≥18 years at the time the ICF is signed (if the legal age of consent is > 18 years old, then follow the local regulatory requirements).
* Histologically or cytologically confirmed unresectable locally advanced (T4b, any N; or any T, N 2-3) or metastatic (any T, any N, M1) urothelial carcinoma of the bladder, renal pelvis, ureter, or urethra.

Participants with urothelial carcinoma (transitional cell) with squamous differentiation or mixed cell types are eligible if the histology is predominantly urothelial.

* Note 1: Urachal, small cell, and adenocarcinoma histology is not permitted.
* Note 2: Participants with la/mUC and a history of nonclinically active prostate cancer are allowed into the trial if:

  1. Participant does not have radiological metastasis of a proven prostate cancer.
  2. Participant with nonmetastatic prostate cancer do not have rising PSA (as determined using local testing by a validated or approved test method) defined as follows:

     • Increase in PSA within 2 consecutive measurements separated by at least 1 week (completed within 4 weeks prior to consent or within Screening) and neither of the measurements with an absolute value above 2 ng/mL.
  3. Participant does not currently receive androgen deprivation therapy for the treatment of prostate cancer. • Must provide tumor tissue sample from archival tissue or newly obtained pretreatment biopsy for exploratory biomarker testing. Tumor tissue sample should not be collected from a lesion that was irradiated unless documentation can be provided confirming that the tumor tissue was collected at least 3 months after radiation and the lesion increased/appeared since radiation occurred. Tumor tissue must be of sufficient quantity (as defined in the laboratory manual).

  <!-- -->

  1. Archival tissue collected after the most recent anticancer treatment and within 12 months before the informed consent date is preferred. • Participant must be considered eligible to receive cisplatin- or carboplatin-containing chemotherapy, in the investigator's judgment. Participants eligible for cisplatin will receive cisplatin. If a participant received gemcitabine, carboplatin or cisplatin for early UC in the adjuvant/neoadjuvant setting, ≥1 year must have passed since the last dose of these chemotherapy prior to the first dose of trial intervention. Participants only receive carboplatin if they are ineligible for cisplatin. Participants are cisplatin-ineligible if they meet any of the following criteria:

  <!-- -->

  1. GFR <60 mL/min (GFR may be estimated by calculated CrCl using the Cockcroft-Gault formula, Modification of Diet in Renal Disease, or 24-hour urine)

     * Participants with a GFR <60 mL/min but ≥50 mL/min but have no other cisplatin ineligibility criteria (items b, c, and d) may be considered cisplatin-eligible based on the investigator's clinical judgment.
  2. NCI-CTCAE Grade ≥2 audiometric hearing loss
  3. NCI-CTCAE Grade ≥2 peripheral neuropathy
  4. NYHA Class III heart failure • Must have experienced radiographic progression or relapse during or after 1L of EV and pembrolizumab.

Participant who discontinued EV and pembrolizumab in 1L due to toxicity are eligible if they have experienced disease progression following discontinuation. Participant who received EV (or other agents with a vedotin payload) plus PD 1/PD-L1 inhibitors in a neoadjuvant/adjuvant setting and progressed during treatment or within 12 months of treatment completion will also be considered for enrollment, after approval by the Sponsor's Medical Monitor or Sponsor's designee.

Key Exclusion Criteria:

* Has had prior systemic therapy other than the combination of EV and pembrolizumab for la/mUC. The following participants may be considered eligible after approval by the Sponsor's Medical Monitor or Sponsor's designee.

  a. Participant who progressed during or after treatments with assets that include either anti-Nectin 4 or vedotin payload (MMAE or other microtubule inhibitors) combined with PD1/PD-L1 inhibitors in 1L la/mUC.
* Treatment with any of the following:

  1. History of an allogeneic bone marrow or solid organ transplant.
  2. Concomitant treatment with any prohibited medications in this protocol.
  3. Prior TROP2 directed ADC therapy.
* Uncontrolled or significant cardiovascular disease, including:

  1. QTcF interval >450 ms based on the average of triplicate 12-lead (ECG per local read) at Screening.
  2. Myocardial infarction within 6 months prior to randomization.
  3. Uncontrolled angina pectoris within 6 months prior to randomization.
  4. NYHA Class 3 or 4 congestive heart failure at Screening (See Section 10.3.2).
  5. Uncontrolled hypertension (resting systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg within 28 days before randomization that is not resolved despite maximal medical therapy).
* Has a history of non-infectious ILD/pneumonitis including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at Screening.
* Has clinically severe pulmonary compromise as judged by the investigator resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (eg, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.) or any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc.), or prior complete pneumonectomy.
* Toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet improved to NCI-CTCAE version 5.0 Grade ≤1 or baseline. Note: Participants may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to Grade >2 for at least 3 months prior to randomization and managed with standard of care treatment) which the investigator deems related to previous anticancer therapy, comprised of (including but not limited to):

  1. Anticancer therapy-induced neuropathy
  2. Residual toxicities from prior immunotherapy treatment: Grade 1 or Grade 2 endocrinopathies which may include:
* Hypothyroidism/ hyperthyroidism
* Type I diabetes
* Hyperglycemia
* Adrenal insufficiency
* Adrenalitis c. Skin hypopigmentation (vitiligo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-01-22 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate - Part A (Phase 2) | From Phase 2 randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, up to approximately 34 months
  Overall Response Rate (ORR) is defined as the proportion of participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or confirmed Partial Response (PR). As assessed by investigator per RECIST v1.1
Progression Free Survival as Assessed by Blinded Independent Central Review (BICR) - Part B (Phase 3) | From Phase 3 randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, up to approximately 38 months
  Progression Free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first. As assessed by BICR per RECIST v1.1
Overall Survival - Part B (Phase 3) | From Phase 3 randomization to death due to any cause, up to approximately 38 months
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Duration of Response - Part A (Phase 2) | From the date of first documentation of objective tumor response to the date of the first documented radiographic disease progression or death due to any cause, whichever occurs first in Phase 2, up to approximately 34 months
  Duration of Response (DoR) is defined as the time from the date of first documentation of objective tumor response (confirmed CR or confirmed PR) to the date of the first documented radiographic disease progression or death due to any cause, whichever occurs first in responding participants. As assessed by investigator per RECIST v1.1
Progression Free Survival as Assessed by Investigator - Part B (Phase 3) | From Phase 3 randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, up to approximately 38 months
  PFS is defined as the time interval from the date of randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first. As assessed by investigator per RECIST v1.1
Overall Response Rate - Part B (Phase 3) | From Phase 3 randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, up to approximately 38 months
  ORR is defined as the proportion of participants with a BOR of confirmed CR or confirmed PR. As assessed by BICR and investigator per RECIST V1.1

CONTACTS AND LOCATIONS:
Locations (64):
- United States (24):
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Aurora, Colorado
  - Research Site, Orange City, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Locust Grove, Georgia
  - Research Site, Effingham, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Largo, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Madison, Wisconsin
- Austria (2):
  - Research Site, Krems
  - Research Site, Vienna
- Umhat 'Sv. Georgi', Ead, Plovdiv, Bulgaria
- China (3):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Guangzhou
- France (19):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Calais
  - Research Site, Cedex 10
  - Research Site, Créteil
  - Research Site, La Chaussée-Saint-Victor
  - Research Site, Le Mans
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Quint-Fonsegrives
  - Research Site, Reims
  - Research Site, Saint-Etienne
  - Research Site, Saint-Herblain
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (2):
  - Universitaetsklinikum Leipzig, Klinik fuer Haematologie, Internistische Onkologie, Haemostaseologische, Leipzig
  - Research Site, Nürtingen
- Italy (2):
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (11):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kawasaki
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Toyama
  - Research Site, Ube-shi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that have reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/